CLINICAL TRIAL: NCT05099003
Title: A Phase 1/2 Trial of Selinexor (KPT-330) and Radiation Therapy in Newly-Diagnosed Pediatric Diffuse Intrinsic Pontine Glioma (DIPG) and High-Grade Glioma (HGG)
Brief Title: A Study of the Drug Selinexor With Radiation Therapy in Patients With Newly-Diagnosed Diffuse Intrinsic Pontine (DIPG) Glioma and High-Grade Glioma (HGG)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-11337; NCI-2021-11337 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS1821 (Other: Children's Oncology Group); ACNS1821 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2021-10-28; First posted 2021-10-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — Biopsy; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (selinexor and radiation therapy) (Experimental): CHEMORADIOTHERAPY: Patients receive standard of care radiation therapy 5 days per week for 5-7 weeks. Starting on day 4 or 5 of radiation therapy, patients receive selinexor PO on 1, 8, 15, 22, 29, 36, 43, and 50 in the absence of disease progression or unacceptable toxicity. After a 2-week rest period, patients proceed to Maintenance. Patients undergo a MRI and may undergo a biopsy during screening.
  MAINTENANCE: Patients receive selinexor PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for up to 24 cycles of maintenance therapy in the absence of disease progression or unacceptable toxicity. Patients undergo a MRI on study and during follow-up.
  Interventions: Procedure: Biopsy Procedure; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Drug: Selinexor

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo a biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Magnetic Resonance Imaging — Undergo a MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Selinexor — Given orally
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT 330; KPT-330; KPT330; Nexpovio; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio

SUMMARY:
This phase I/II trial tests the safety, side effects, and best dose of selinexor given in combination with standard radiation therapy in treating children and young adults with newly diagnosed diffuse intrinsic pontine glioma (DIPG) or high-grade glioma (HGG) with a genetic change called H3 K27M mutation. It also tests whether combination of selinexor and standard radiation therapy works to shrink tumors in this patient population. Glioma is a type of cancer that occurs in the brain or spine. Glioma is considered high risk (or high-grade) when it is growing and spreading quickly. The term, risk, refers to the chance of the cancer coming back after treatment. DIPG is a subtype of HGG that grows in the pons (a part of the brainstem that controls functions like breathing, swallowing, speaking, and eye movements). This trial has two parts. The only difference in treatment between the two parts is that some subjects treated in Part 1 may receive a different dose of selinexor than the subjects treated in Part 2. In Part 1 (also called the Dose-Finding Phase), investigators want to determine the dose of selinexor that can be given without causing side effects that are too severe. This dose is called the maximum tolerated dose (MTD). In Part 2 (also called the Efficacy Phase), investigators want to find out how effective the MTD of selinexor is against HGG or DIPG. Selinexor blocks a protein called CRM1, which may help keep cancer cells from growing and may kill them. It is a type of small molecule inhibitor called selective inhibitors of nuclear export (SINE). Radiation therapy uses high energy to kill tumor cells and shrink tumors. The combination of selinexor and radiation therapy may be effective in treating patients with newly-diagnosed DIPG and H3 K27M-Mutant HGG.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define toxicities and estimate the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of selinexor administered as an oral formulation in combination with standard of care radiation therapy (RT), to pediatric patients with newly diagnosed high-grade glioma (HGG) or diffuse intrinsic pontine glioma (DIPG). (Dose-finding phase/phase I) II. To estimate the event-free survival (EFS) distribution for diffuse midline glioma (DMG)/HGG patients and overall survival (OS) distribution for DIPG patients associated with selinexor plus RT, followed by selinexor in patients with newly diagnosed HGG (H3 K27M mutant DMG or H3 K27-wild type HGG) or DIPG, and to compare those outcomes to historical controls. (Efficacy phase/phase II)

EXPLORATORY OBJECTIVE:

I. To bank tumor specimens and body fluids (blood and cerebrospinal fluid) for future studies.

OUTLINE: This is a phase I dose-escalation study of selinexor followed by a phase II study. (STRATUM DIPG AND STRATUM DMG CLOSED TO ACCRUAL 02/14/2025)

CHEMORADIOTHERAPY: Patients receive standard of care radiation therapy 5 days per week for 5-7 weeks. Starting on day 4 or 5 of radiation therapy, patients receive selinexor orally (PO) on days 1, 8, 15, 22, 29, 36, 43, and 50 in the absence of disease progression or unacceptable toxicity. After a 2-week rest period, patients proceed to Maintenance. Patients undergo a magnetic resonance imaging (MRI) and may undergo a biopsy during screening.

MAINTENANCE: Patients receive selinexor PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for up to 24 cycles of maintenance therapy in the absence of disease progression or unacceptable toxicity. Patients undergo a MRI on study and during follow-up.

After completion of study treatment, patients are followed every 3 months for year 1 (i.e., 3, 6, 9, 12 months), then every 6 months for years 2-3 (i.e., 18, 24, 30, 36 months), and finally once yearly for years 4-5 of this study.

ELIGIBILITY:
Inclusion Criteria:

* PRE ENROLLMENT: Patients must be =< 25 years of age at the time of enrollment on APEC14B1 part A central nervous system (CNS)/high grade glioma (HGG) pre-enrollment eligibility screening

  * Please note:

    * This required age range applies to pre-enrollment eligibility for all HGG patients. Individual treatment protocols may have different age criteria.
    * Non-DIPG patients with tumors that do not harbor an H3K27M-mutation and are >= 18 years of age will not be eligible to enroll on ACNS1821 (Step 1).
* PRE ENROLLMENT: Patient is suspected of having localized, newly diagnosed HGG, excluding metastatic disease, OR patient has an institutional diagnosis of DIPG

  * Please note: there are specific radiographic criteria for DIPG patient enrollment on ACNS1821 (Step 1)
  * As of February 14, 2025, stratum DIPG and stratum DMG have closed to accrual, and no patients will be enrolled on these strata after Amendment #4.
* PRE ENROLLMENT:

  * For patients with non-pontine tumors: Patients and/or their parents or legal guardians must have signed informed consent for eligibility screening on APEC14B1 Part A.
  * For patients with DIPG: Patients and/or their parents or legal guardians must have signed informed consent for ACNS1821.
  * Note: As of February 14, 2025, stratum DIPG and stratum DMG have closed to accrual, and no patients will be enrolled on these strata after Amendment #4.
* PRE ENROLLMENT:

  * For patients with non-pontine tumors only, the specimens obtained at the time of diagnostic biopsy or surgery must be submitted through APEC14B1 ASAP, preferably within 5 calendar days of definitive surgery
* STEP 1: Patients must be >= 12 months and =< 21 years of age at the time of enrollment
* STEP 1: Patients must have newly-diagnosed DIPG or HGG (including DMG).
* STEP 1: Stratum DIPG (Closed with Amendment #4)

  * As of February 14, 2025, stratum DIPG and stratum DMG have closed to accrual, and no patients will be enrolled on these strata after Amendment #4.
  * Patients with newly-diagnosed typical DIPG, defined as tumors with a pontine epicenter and diffuse involvement of at least 2/3 of the pons on at least 1 axial T2 weighted image, are eligible. No histologic confirmation is required.
  * Patients with pontine tumors that do not meet radiographic criteria for typical DIPG (e.g., focal tumors or those involving less than 2/3 of the pontine cross-sectional area with or without extrapontine extension) are eligible if the tumors are biopsied and proven to be high-grade gliomas (such as anaplastic astrocytoma, glioblastoma, high-grade glioma not otherwise specified [NOS], and/or H3 K27M-mutant) by institutional diagnosis.
* STEP 1: Stratum DMG (with H3 K27M mutation) (Closed with Amendment #4)

  * As of February 14, 2025, stratum DIPG and stratum DMG have closed to accrual, and no patients will be enrolled on these strata after Amendment #4.
  * Patients must have newly-diagnosed non-pontine H3 K27M-mutant HGG without BRAF V600 or IDH1 mutations as confirmed by Rapid Central Pathology and Molecular Screening Reviews performed on APEC14B1
  * Note: Patients need not have either measurable or evaluable disease, i.e., DMG patients may have complete resection of their tumor prior to enrollment. Primary spinal tumors are eligible for enrollment. For rare H3 K27M-mutant HGG in non-midline structures (e.g., cerebral hemispheres), these patients will be considered part of Stratum DMG.
* STEP 1: Stratum HGG (without H3 K27M mutation)

  * Patients must have newly-diagnosed non-pontine H3 K27M-wild type HGG without BRAF V600 or IDH1 mutations as confirmed by Rapid Central Pathology and Molecular Screening Reviews performed on APEC14B1
  * Please note:

    * Patients who fall in this category and who are >= 18 years of age are not eligible due to another standard-of-care regimen (radiation/temozolomide) that is available
    * Patients need not have either measurable or evaluable disease, i.e., HGG patients may have complete resection of their tumor prior to enrollment. Primary spinal tumors are eligible for enrollment
* STEP 1: Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =<16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* STEP 1: Peripheral absolute neutrophil count (ANC) >= 1000/uL (within 7 days prior to step 1 enrollment)
* STEP 1: Platelet count >= 100,000/uL (transfusion independent) (within 7 days prior to step 1 enrollment)
* STEP 1: Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions) (within 7 days prior to step 1 enrollment)
* STEP 1: Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 (within 7 days prior to step 1 enrollment) or

A serum creatinine based on age/sex as follows (within 7 days prior to step 1 enrollment):

* Age / Maximum Serum Creatinine (mg/dL)

  * 1 to < 2 years / male: 0.6; female: 0.6
  * 2 to < 6 years / male: 0.8; female: 0.8
  * 6 to < 10 years / male: 1; female: 1
  * 10 to < 13 years / male: 1.2; female: 1.2
  * 13 to < 16 years / male: 1.5; female: 1.4
  * >= 16 years / male: 1.7; female: 1.4

    * STEP 1: Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
    * STEP 1: Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
    * STEP 1: Serum amylase =< 1.5 x ULN
    * STEP 1: Serum lipase =< 1.5 x ULN
    * STEP 1: No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination.
    * STEP 1: Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled.
    * STEP 1: Patients must be enrolled and protocol therapy must begin no later than 31 days after the date of radiographic diagnosis (in the case of non-biopsied DIPG patients only) or definitive surgery, whichever is the later date (Day 0).

For patients who have a biopsy followed by resection, the date of resection will be considered the date of definitive diagnostic surgery. If a biopsy only was performed, the biopsy date will be considered the date of definitive diagnostic surgery.

Exclusion Criteria:

* STEP 1: Patients must not have received any prior therapy for their central nervous system (CNS) malignancy except for surgery and steroid medications.
* STEP 1: Patients who are currently receiving another investigational drug are not eligible.
* STEP 1: Patients who are currently receiving other anti-cancer agents are not eligible.
* STEP 1: Patients >=18 years of age who have H3 K27M-wild type HGG.
* STEP 1: Patients who have an uncontrolled infection.
* STEP 1: Patients who have received a prior solid organ transplantation.
* STEP 1: Patients with grade > 1 extrapyramidal movement disorder.
* STEP 1: Patients with known macular degeneration, uncontrolled glaucoma, or cataracts.
* STEP 1: Patients with metastatic disease are not eligible; MRI of spine with and without contrast must be performed if metastatic disease is suspected by the treating physician.
* STEP 1: Patients with gliomatosis cerebri type 1 or 2 are not eligible, with the exception of H3 K27M-mutant bithalamic tumors.
* STEP 1: Patients who are not able to receive protocol specified radiation therapy.
* STEP 1:

  * Female patients who are pregnant are ineligible since there is yet no available information regarding human fetal or teratogenic toxicities.
  * Lactating females are not eligible unless they have agreed not to breastfeed their infants. It is not known whether selinexor is excreted in human milk.
  * Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained.
  * Sexually active patients of reproductive potential are not eligible unless they have agreed to use two effective methods of birth control (including a medically accepted barrier method of contraception, e.g., male or female condom) for the duration of their study participation and for 90 days after the last dose of selinexor. Abstinence is an acceptable method of birth control.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | From day 1 of selinexor treatment until the start of maintenance therapy, assessed up to 10 weeks from treatment start date
  Defined as the highest dose of selinexor in combination with standard of care radiation therapy (RT) that does not cause unacceptable side effects.
Event free survival (EFS) | From the date of enrollment until disease progression date, secondary malignant neoplasm occurrence date, death date of any cause, or last follow-up date, assessed up to 5 years
  Will be calculated for diffuse midline glioma (DMG)/ high grade glioma (HGG) patients. EFS curve will be estimated by Kaplan Meier estimates.
Overall Survival (OS) | From the date of enrollment until death date of any cause or last follow-up date, assessed up to 5 years
  Will be calculated for diffuse intrinsic pontine glioma (DIPG) patients. The OS curve will be estimated by Kaplan Meier estimates.
Overall response rate (ORR) | Up to 5 years
  Defined as the proportion of patients whose best response is partial response or complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Adam L Green, Principal Investigator — Children's Oncology Group
Locations (127):
- United States (109):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm